CLINICAL TRIAL: NCT00005177
Title: Reno Diet Heart Study
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1055; R01HL034589 (NIH)
Record Dates: First submitted 2000-05-25; First posted 2000-05-26 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2000-06

CONDITIONS: Cardiovascular Diseases; Heart Diseases; Obesity
MeSH Terms: conditions — Cardiovascular Diseases; Heart Diseases; Obesity

SUMMARY:
To study weight maintenance behaviors, weight trends, and behavioral differences between healthy, normal weight and mildly obese adults.

DETAILED DESCRIPTION:
BACKGROUND:

The treatment of obesity has met with limited success and clinically significant weight losses have been difficult to achieve and maintain. Screening to determine which patient will benefit most from treatment, emphasis on maintenance of weight loss and understanding individual weight trends and goals, all have demonstrated significant impact on long-term treatment outcome. Stunkard established a new classification of obesity according to severity and predicted outcome to treatment, distinguishing mild and moderate overweight from severe forms of obesity. Those who were classified as mildly obese were those who were most likely to be successful in traditional forms of treatment. A comprehensive study of this mildly obese population and normal weight maintenance behaviors provided important information on which to build future treatment interventions and/or effective strategies. This would be of particular importance in the prevention of obesity and progressive escalation of the obese state.

DESIGN NARRATIVE:

Subjects were studied retrospectively by history and prospectively in their natural setting for five years. A 2 x 2 x 5 multifactorial design was used where sex (males versus females) and weight (obese versus normal) were crossed with five different age groups according to decades (20-29, 30-39, 40-49, 50-59 and 60 or more years) respectively. A total of 50 (25 normal and 25 obese) were recruited for each age/sex group. Dependent variables included: weight, weight trends, fluctuation, body composition; diet; activity or exercise; weight maintenance behaviors and adaptive responses; general well-being, emotional states, psychopathology; routine blood and urinalyses; cardiovascular disease risk profile including lipids, blood pressure, sodium, potassium, calcium and phosphorus levels, diet, smoking, alcohol and caffeine use, onset of menopause and changes in medical status or medication use. Comprehensive assessment was done yearly.

The study was renewed in 1992 to extend follow-up and evaluation of the RENO Diet Heart Study and to complete and extend testing of the primary hypotheses. The three major hypotheses tested included: 1) weight fluctuations affected cardiovascular disease (CVD) risk factors over and above weight change alone; 2) weight changes, fluctuations and patterns interacted with nutritional, behavioral, psychological and medical factors, but these factors also affected CVD risk independent of weight; and 3) retrospective, self-reported weights, fluctuations and patterns were predictive of prospective weights and weight fluctuations.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1985-09; Study Completion 1996-11 (Actual)

REFERENCES:
- [Background] St. Jeor ST, Sutnik M, Scott B: Nutrition. In: Behavioral Medicine for Women. Bleckman EA, Brownell KD (Eds), Elmsford, NY: Permagon Press, 1987
- [Background] Read MA, Brunner RL, Miller G, St Jeor ST, Scott BJ, Carmody TP. Relationship of vitamin/mineral supplementation to certain psychologic factors. J Am Diet Assoc. 1991 Nov;91(11):1429-31. No abstract available. PMID 1939983
- [Background] Mifflin MD, St Jeor ST, Hill LA, Scott BJ, Daugherty SA, Koh YO. A new predictive equation for resting energy expenditure in healthy individuals. Am J Clin Nutr. 1990 Feb;51(2):241-7. doi: 10.1093/ajcn/51.2.241. PMID 2305711
- [Background] Foreyt JP, Brunner RL, Goodrick GK, St Jeor ST, Miller GD. Psychological correlates of reported physical activity in normal-weight and obese adults: the Reno diet-heart study. Int J Obes Relat Metab Disord. 1995 Oct;19 Suppl 4:S69-72. PMID 8581099
- [Background] Carmody TP, Brunner RL, St Jeor ST. Dietary helplessness and disinhibition in weight cyclers and maintainers. Int J Eat Disord. 1995 Nov;18(3):247-56. doi: 10.1002/1098-108x(199511)18:33.0.co;2-w. PMID 8556020
- [Background] Foreyt JP, Brunner RL, Goodrick GK, Cutter G, Brownell KD, St Jeor ST. Psychological correlates of weight fluctuation. Int J Eat Disord. 1995 Apr;17(3):263-75. doi: 10.1002/1098-108x(199504)17:33.0.co;2-n. PMID 7773263
- [Background] Katz DL, Brunner RL, St Jeor ST, Scott B, Jekel JF, Brownell KD. Dietary fat consumption in a cohort of American adults, 1985-1991: covariates, secular trends, and compliance with guidelines. Am J Health Promot. 1998 Jul-Aug;12(6):382-90. doi: 10.4278/0890-1171-12.6.382. PMID 10182090
- [Background] St Jeor ST, Brunner RL, Harrington ME, Scott BJ, Daugherty SA, Cutter GR, Brownell KD, Dyer AR, Foreyt JP. A classification system to evaluate weight maintainers, gainers, and losers. J Am Diet Assoc. 1997 May;97(5):481-8. doi: 10.1016/S0002-8223(97)00126-0. PMID 9145085
- [Background] St Jeor ST, Brunner RL, Harrington ME, Scott BJ, Cutter GR, Brownell KD, Dyer AR, Foreyt JP. Who are the weight maintainers? Obes Res. 1995 Sep;3 Suppl 2:249s-259s. doi: 10.1002/j.1550-8528.1995.tb00471.x. PMID 8581784